CLINICAL TRIAL: NCT02419183
Title: A Randomized Cross-over, Controlled Feasibility, and Validation Study of a Self-Administered Memory Screening Test With Automated Reporting (SAMSTAR) in Subjects With Mild Cognitive Impairment
Brief Title: A Study of a Self-Administered Memory Screening Test With Automated Reporting (SAMSTAR) in Participants With Mild Cognitive Impairment
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR106702; NOPRODALZ0001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Self-Administered Memory Screening Test With Automated Reporting (SAMSTAR); Rey Auditory Verbal Learning Test (RAVLT); Word List Recall (WLR)
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sequence A: Participants will receive a computer administered Word List Recall (WLR) [SAMSTAR] on Test Day 1 and an examiner addminstered WLR [RAVLT] on Test Day 2 of the study.
  Interventions: Other: SAMSTAR; Other: RAVLT
- Sequence B: Participants will receive an examiner-administered WLR [RAVLT] on Test Day 1 and a computer adminstered WLR [SAMSTAR] on Test Day 2 of the study.
  Interventions: Other: SAMSTAR; Other: RAVLT

INTERVENTIONS:
Other: SAMSTAR — This is a non-interventional study based on computer-administered WLR (SAMSTAR) test and examiner-administered WLR (RAVLT) test to investigate whether the performance of participants is equivalent.
Other: RAVLT — This is a non-interventional study based on computer-administered WLR (SAMSTAR) test and examiner-administered WLR (RAVLT) test to investigate whether the performance of participants is equivalent.

SUMMARY:
The purpose of this study is to evaluate the psychometric properties of a Self-administered Memory Screening Test with Automated Reporting (SAMSTAR) adapted from the Rey Auditory Verbal Learning Test (RAVLT) in normal control (NC) participants and participants with Mild Cognitive Impairment (MCI) against a standard version of the RAVLT test, administered by an examiner under the same conditions.

DETAILED DESCRIPTION:
This is a single-center (when only one hospital or medical school team work on a medical research study), randomized (participants are assigned to treatment by a chance), crossover (participants may receive different treatments sequentially during the trial) study. The study consists of a Screening Phase (Day -3 up to and including Day 1), Test Phase (Test Day 1 and Test Day 2 [within 7 to 14 days following Test Day 1]) and an optional follow-up visit within 7 days after the last study-related activity for participants who experienced an adverse event that had not resolved by the end of the last test visit.The NC and MCI participants will initially either undergo a standard version of the RAVLT test or the SAMSTAR version of the RAVLT test on Test Day 1 or on the same day as screening, with follow-up testing using the other test using a crossover design to be conducted within 1 to 2 weeks at the same venue (Test Day 2). There will be a 7-to 14-day memory washout period between the test periods. No investigational medicinal product will be administered. The maximum study duration for a participant will not exceed 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have normal visual and hearing acuity (corrected or uncorrected) as assessed in the Screening cognitive test (MoCA)
* Screening Criteria:

  1. NC participants: meet inclusion/exclusion criteria, Dementia Screening Interview (8- item) (AD8) score 0-1, MoCA score 28 or higher (education-adjusted)
  2. MCI participants: meet inclusion/exclusion criteria, AD8 score 2 or higher, MoCA score 24 to 27 (education-adjusted)
* Participant must be English-speaking and able to understand and follow the examiner/trial instructions
* Each participant must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Participant has an acute or chronic medical condition (eg, Alzheimer's disease [AD] or depression) that would interfere with the participant's ability to complete either memory test assessment or comply with other study requirements
* Participant has an acute or chronic psychiatric condition that would interfere with the participant's ability to complete either memory test assessment or comply with other study requirements
* Participant has any acute or chronic neurological conditions (eg, stroke, epilepsy, Parkinson's disease)
* Participant has any sensory, motor or speech impairment that would interfere with the participants' ability to complete memory testing that relies on speech recognition
* Participant has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Ages: 55 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female adult normal control (NC) participants and participants with Mild Cognitive Impairment (MCI), aged 55 to 84 years receiving healthcare in primary care and/or neurology practice settings.
Sampling Method: Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Cognitive Evaluation by Self-administered memory screening test with automated reporting (SAMSTAR) | Up to 3 weeks
  The memory test will include a list of 15 words presented one at a time through the iPad (on screen and aloud). After the 15-word list is presented, the participant will be asked to verbally recall as many of the words as possible.
Cognitive Evaluation by Rey Auditory Verbal Learning Test (RAVLT) | Up to 3 weeks
  The memory test will include a list of 15 words presented one at a time verbally by the examiner. After the 15-word list is presented, the participant will be asked to verbally recall as many of the words as possible.

SECONDARY OUTCOMES:
Assess the feasibility of SAMSTAR | Up to 3 weeks
  The feasibility of using a SAMSTAR approach to cognitive screening will be evaluated by meeting target enrollment criteria and by survey data from participants and clinical staff about their experience and attitudes regarding cognitive screening as executed in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- United States (2):
  - Chapel Hill, North Carolina
  - Durham, North Carolina